CLINICAL TRIAL: NCT07405073
Title: Advanced Practice Nurse Specializing in Emergency and Post-emergency Care: Towards Improved Unscheduled Care?
Brief Title: Advanced Practice Nurse Specializing in Emergency Care and Post-emergency Consultation: Feasibility Study
Acronym: CPU - IPA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-05-Obs-CHRMT
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Healthcare Access

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Emergency departments are facing increasing overload, exacerbated by difficulties in accessing primary care. This saturation impacts the fluidity of care pathways and the quality of care.

A major challenge is the high rate of short-term repeat visits, which increases the workload. These early returns may be due to an unexpected change in the patient's condition, but also to the difficulty of obtaining a quick appointment with a general practitioner, due to a shortage of practitioners or a lack of available slots within a few days.

DETAILED DESCRIPTION:
In this context, the implementation of a Post-Emergency Consultation by an Advanced Practice Nurse could be a solution to improve patient follow-up and limit these avoidable return visits.

Main objective: Identify the profiles of patients who return for a second consultation within 15 days of their first visit to the emergency department.

Secondary objectives:

* Describe the characteristics of these patients (age, gender, medical history, pathologies, reasons for the initial consultation, reasons for the repeat consultation).
* Analyze medical records to assess whether a post-emergency consultation by an APN could have prevented this repeat consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visited the emergency department at 15-day intervals during the study period

Exclusion Criteria:

* Patients hospitalized at the time of the first consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited the emergency department and were seen again within 15 days.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage patients who return for a second consultation | 15 days
  Percentage of patients who return for a second consultation within 15 days of their first visit to the emergency department and prifile of patients

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No